CLINICAL TRIAL: NCT03005106
Title: A Phase III Open-label, Controlled, Randomized, Multicenter Study Evaluating the Efficacy and Safety of StrataGraft Skin Tissue in Promoting Autologous Skin Tissue Regeneration of Complex Skin Defects Due to Thermal Burns That Contain Intact Dermal Elements and for Which Excision and Autografts Are Clinically Indicated
Brief Title: StrataGraft® Skin Tissue in the Promotion of Autologous Skin Regeneration of Complex Skin Defects Due to Thermal Burns That Contain Intact Dermal Elements
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRATA2016
Expanded Access: Available
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Burn, Thermal
Keywords: Trauma-related wound; Deep partial thickness; Skin wound
MeSH Terms: conditions — Burns | interventions — Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: See detailed description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- StrataGraft Skin Tissue (Experimental)
  Interventions: Biological: StrataGraft Skin Tissue; Procedure: Autograft

INTERVENTIONS:
Biological: StrataGraft Skin Tissue — StrataGraft® skin tissue is provided as a suturable rectangular piece of stratified epithelial tissue composed of a living dermal matrix containing dermal fibroblasts overlaid with human epidermal keratinocytes (NIKS®).
Procedure: Autograft — The current standard of care procedure for the treatment of severe burns. The procedure involves the removal of a sheet of healthy skin from an uninjured site on the patient and using it to cover the original burn wound.

SUMMARY:
About 70 participants will be enrolled. They will have complex skin defects because of burns caused by heat.

The burns will:

* be on 3-49% of the participant's total body surface area (TBSA)
* require surgery for skin replacement
* include intact dermal elements

The burns are called deep, partial-thickness thermal burns because the skin was damaged by heat but still has some dermis that was not damaged.

The dermis is the layer of skin under the outer layer (epidermis). It is the thickest layer of the skin that provides strength and flexibility to the skin.

All patients will receive both treatments, but on different areas of their burns. Their wounds will not be compared to other patients. One treatment area on their own body will be compared to the other one.

This will help to find out if StrataGraft is safe and effective for deep partial thickness burns. It will also see if StrataGraft might help healing enough to use it instead of the patient's own healthy skin to repair the damage.

ELIGIBILITY:
Inclusion Criteria

Subject-specific criteria:

1. Men and women aged ≥ 18 years
2. Written informed consent
3. Sufficient healthy skin identified and reserved as a donor site in the event that the StrataGraft treatment site requires autografting
4. Clinical expectation that the study donor site will heal without grafting
5. Complex skin defects of 3-49% TBSA

   * Total burn may consist of more than one area

   Treatment site-specific criteria:
6. Thermal burn(s) with intact dermal elements for which excision and autografting are clinically indicated
7. Total of both study treatment areas can be up to 2000 cm2
8. First excision and grafting of study treatment sites
9. Thermal burn(s) on the torso, arms, or legs

Exclusion Criteria

Subject-specific criteria:

1. Pregnant women
2. Prisoners
3. Subjects receiving systemic immunosuppressive therapy
4. Subjects with a known history of malignancy
5. Preadmission insulin-dependent diabetic subjects
6. Subjects with concurrent conditions that in the opinion of the investigator may compromise subject safety or study objectives
7. Expected survival of less than three months
8. Participation in the treatment group of an interventional study within 90 days prior to enrollment

   Treatment site-specific criteria:
9. Full-thickness burns
10. Chronic wounds
11. The face, head, neck, hands, feet, buttocks, and area over joints
12. Treatment sites immediately adjacent to unexcised eschar
13. Clinical or laboratory determination of infection at the anticipated treatment sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Stratatech, a Mallinckrodt Company
Locations (16):
- United States (16):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Arizona Burn Center at Maricopa Medical Center, Phoenix, Arizona
  - Universtiy of California - Irvine Health Regional Burn Center, Orange, California
  - UC Davis, Sacramento, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Health Shands Burn Center, Gainesville, Florida
  - Tampa General Hospital - Regional Burn Center, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Baton Rouge Medical Center, Baton Rouge, Louisiana
  - University Medical Center, New Orleans, Louisiana
  - University of Missouri, Columbia, Missouri
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Regional Medical Center Firefighters Burn Center, Memphis, Tennessee
  - U.S. Army Institute of Surgical Research Adult Burn Center, Fort Sam Houston, Texas
  - University of Wisconsin Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT03005106) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Gibson ALF, Holmes JH 4th, Shupp JW, Smith D, Joe V, Carson J, Litt J, Kahn S, Short T, Cancio L, Rizzo J, Carter JE, Foster K, Lokuta MA, Comer AR, Smiell JM, Allen-Hoffmann BL. A phase 3, open-label, controlled, randomized, multicenter trial evaluating the efficacy and safety of StrataGraft(R) construct in patients with deep partial-thickness thermal burns. Burns. 2021 Aug;47(5):1024-1037. doi: 10.1016/j.burns.2021.04.021. Epub 2021 Apr 23. PMID 34099322

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: StrataGraft Skin Tissue: StrataGraft® skin tissue is provided as a suturable rectangular piece of stratified epithelial tissue composed of a living dermal matrix containing dermal fibroblasts overlaid with human epidermal keratinocytes (NIKS®).
  Autograft: The current standard of care procedure for the treatment of severe burns. The procedure involves the removal of a sheet of healthy skin from an uninjured site on the patient and using it to cover the original burn wound.
Period: Overall Study
Arm/Group | All Participants
Started | 71
Completed Month 3 Visit | 64
Completed Month 12 Visit | 51
Completed | 51
Not Completed | 20
Not completed — Lost to Follow-up | 16
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 55
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Percent Area of Treatment Sites Requiring Autografting by Month 3
Description: Percent area autografted by Month 3 is the sum of the percent areas at each study session/visit, up to and including Study Session 7/Month 3 (± 14 d).
Time Frame: 3 Months
Population: Modified Intent to Treat Population
Measure: Mean (Standard Deviation); unit: percentage of treatment sites
Arm/Group | All Participants
Number analyzed (Participants) | 71
percentage of treatment sites
  StrataGraft (Treatment) Sites | 4.33 (21.58)
  Autograft (Control) Sites | 102.10 (13.14)
Statistical Analysis 1: Comparison: All Participants; Test type: Other — Difference between treatment and control sites; p < 0.0001, one-sided Wilcoxin Signed RankTtest — Difference is (percent area of Autograft treatment site requiring autografting by Month 3) - (percent area of StrataGraft treatment site requiring autografting by Month 3); Mean Difference (Final Values) = 97.77

2. Primary Outcome: Number of Participants Classified as a Responder (Based on Durable Wound Closure at Month 3)
Description: Wound closure of the treatment site was defined as complete skin re-epithelialization and the absence of drainage. A participant whose StrataGraft treatment site achieves durable wound closure without autograft placement is classified as a responder.
Time Frame: Month 3
Population: Modified Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Participants | 59
Statistical Analysis 1: Comparison: All Participants; Test type: Other; Percentage of participants = 83.1, 95% CI 2-sided [74.4 to 91.8] — 95% confidence interval is derived using the normal approximation to the binomial distribution

3. Secondary Outcome: Pain at the Designated Donor Sites by Day 14
Description: Pain scores from the FACES scale range from 0 (no pain) to 5 (worst pain). Pain scores from Day 3, Day 7, and Day 14 (where available) are averaged for the summary statistics.
Time Frame: Day 3, Day 7 and Day 14, average of the 3 days reported
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 71
score on a scale
  StrataGraft (Treatment) | 0.15 (0.54)
  Autograft (Control) | 2.55 (1.30)
Statistical Analysis 1: Comparison: All Participants; Test type: Other — Difference is Autograft - StrataGraft; p < 0.0001, 1-sided, paired t-test; p-value from 1-sided, paired t-test on the mean difference(Autograft - StrataGraft); Mean Difference (Final Values) = 2.40

4. Secondary Outcome: Total Scar Assessment (POSAS) Score by Observer at Month 3
Description: Total Score is the sum of the scores for vascularization, pigmentation, thickness, relief, pliability, and surface area. For each of the 6 assessment categories, the scale ranged from 1=normal skin to 10=worst scar imaginable, with the highest possible score of 10. A higher score indicates worse scarring, so the best possible total score for the 6 categories is 6, and the worst possible score is 60.
Time Frame: at Month 3
Population: Maximum number of participants with data at Month 3 in the modified Intent to Treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 61
score on a scale
  StrataGraft (Treatment) | 6.3 (1.71)
  Autograft (Control) | 16.3 (7.71)
Statistical Analysis 1: Comparison: All Participants; Test type: Other — Difference is Autograft - StrataGraft; p < 0.0001, 1-sided, paired t-test — Missing total score data were imputed using a multiple imputation analysis assuming a monotone missing data pattern. A linear regression model with ethnicity, race and age as predictive variables was used in the imputation; p-value from 1-sided, paired t-test on the difference (Autograft - StrataGraft); Mean Difference (Final Values) = 10.0

ADVERSE EVENTS:
Time Frame: Through the 12-month follow-up
Description: Only Treatment-Emergent Adverse Events (TEAEs) were used for the non-serious adverse events table.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 2/71
Serious Adverse Events (participants affected / at risk) | 10/71
Other Adverse Events (participants affected / at risk) | 49/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=71)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Migraine (Vascular disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Concomitant disease progression (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=71)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 5 (5)
Pain (General disorders) | 8 (8)
Pyrexia (General disorders) | 4 (4)
Donor site complication (Injury, poisoning and procedural complications) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Neuralgia (Nervous system disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 5 (5)
Blister (Skin and subcutaneous tissue disorders) | 10 (12)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 11 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (29)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertension (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT03005106/Prot_SAP_000.pdf